CLINICAL TRIAL: NCT06569888
Title: Utility of Low Intensity Pulsed Ultrasound Stimulation (LIPUS) to Modulate the Release of Mediators Capable of Reflecting the Inflammatory State in the Affected Colonic Tract of Ulcerative Colitis Patients
Acronym: LIPUSinVIVO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Innovative Medicines Initiative (Other); Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IBD-2022-001
Record Dates: First submitted 2024-07-29; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LIPUS stimulation (Experimental): LIPUS stimulation supplying the pre-clinically optimized energy dosage and conditions
  Interventions: Device: LIPUS stimulation

INTERVENTIONS:
Device: LIPUS stimulation — Low Intensity Pulsed Ultrasound stimulation of the gut at the pre-clinically optimized conditions and energy dosage

SUMMARY:
The goal of this clinical trial is to learn whether Low Intensity Pulsed Ultrasound (LIPUS) is capable of promoting the release of extracellular vesicles from the gut into the bloodstream of Ulcerative Colitis (UC) patients, whose content may be predictive of the inflammatory state of the mucosal source to aid the monitoring of the disease status and therapy response.

The main questions it aims to answer are:

Is LIPUS effective in inducing the release of biomarker-containing micro-vesicles into the bloodstream, capable of reflecting the inflammatory state of the mucosa during active disease?

Are there any extracellular vesicle-contained biomarkers that can monitor therapy during clinical remission?

Participants who undergo endoscopy and gut biopsy collection as per Standard Of Care, will:

* undergo abdominal ultrasound to establish the distance with the target tissue and consequently set the LIPUS device to supply the optimum energy established in the protocol.
* before LIPUS stimulation and 2 hours after stimulation, patients will have blood drawn
* an extra intestinal biopsy during endoscopy will be collected
* patients will be contacted 72h after intervention for adverse events monitoring

ELIGIBILITY:
Inclusion Criteria:

For Phase A:

* male and female patients ≥ 18 years of age (at the time of signing the Informed Consent) -signed written Informed Consent
* established diagnosis of UC with a minimum disease duration of 3 months
* moderate, moderate to severe active UC, defined by partial Mayo Score
* indication to start any targeted therapy, yet not initiated
* in case of treatment with corticosteroid: stabile dose for at least 3 weeks prior to baseline, dosage ≤ 20 mg prednisone
* indication for colonoscopy for the assessment of disease activity as for standards of care and current guidelines
* able to comply with the study procedures
* BMI <23.

For Phase B:

* male and female patients ≥ 18 years of age (at the time of signing the Informed Consent)
* signed written Informed Consent
* established diagnosis of UC and in clinical remission defined by partial Mayo Score with any targeted therapy
* able to comply with the study procedures
* BMI <23.

Exclusion Criteria for both phases:

* diagnosis of indeterminate colitis, Crohn's colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis
* absolute contraindications to colonoscopy procedures, complication during previous endoscopy
* bleeding disorders
* indication for surgery for UC
* legal incapacity
* rectal topical therapy (enemas or suppositories) ≤ 2 weeks prior to baseline
* treatment with > 20 mg prednisone within 3 weeks prior to baseline
* anemia (hemoglobin < 10 g/dl) at baseline
* pregnant or breastfeeding women
* women with implanted contraceptive device
* BMI>23
* patients diagnosed with cancer (especially attention goes to colon-rectal neoplasty)
* high turnover osteoporosis
* presence of metal fragments
* joint prostheses
* varicous veins
* phlebitis and thrombophlebitis
* presence of pacemaker
* obliterating arteriopathy
* menstruation
* neoplastic tissues and surrounding areas
* tuberculosis
* individuals in the growing phase (children and adolescents)
* individuals not capable of communicating sense of pain
* any circumstances which could contradict a study participation and lead the Investigator to assess the patient as unsuitable for study participation for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficiency of LIPUS in terms of target-specific extracellular vesicle release | 14 months
  Evaluation of LIPUS efficiency in extracellular vesicle release by measuring extracellular vesicle concentration in blood before and after LIPUS stimulation

SECONDARY OUTCOMES:
Accuracy of LIPUS stimulation in monitoring ulcerative colitis in terms of tissue state-specific biomarkers contained in LIPUS-induced extracellular vesicles | 14 months
  Identification of extracellular vesicle molecular content before and after LIPUS stimulation which correlate with intestinal inflammation in Ulcerative Colitis (active/remission states) by fluorescent miRNA microarray technology and RNA-seq

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Armuzzi, MD, Principal Investigator — Istituto Clinico Humanitas

IPD SHARING:
Plan to Share IPD: No